CLINICAL TRIAL: NCT00775957
Title: Assessment of Hematopoietic Recovery Following Chemotherapy for Non-Hodgknin's Lymphoma
Brief Title: Assessment of Hematopoietic Recovery Following Chemotherapy for Non-Hodgkin's Lymphoma
Status: Terminated | Type: Observational
Why Stopped: Terminated by institutional review board
Sponsor: University of Oklahoma (Other)
Collaborators: Midwest Medical Isotopes (Unknown)
Responsible Party: Jennifer Holter, MD, University of Oklahoma Health Sciences Center- Dept. of Medicine
Other Study IDs: FLT-NHL
Record Dates: First submitted 2008-10-17; First posted 2008-10-20 (Estimated); Last update posted 2010-09-28 (Estimated); Status verified 2010-09

CONDITIONS: Non-Hodgkin's Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: FLT-PET Scan
  Interventions: Procedure: FLT-PET scan
- 2: FDG-PET Scan
  Interventions: Procedure: FDG-PET scan

INTERVENTIONS:
Procedure: FLT-PET scan — imaging scan
  Groups: 1
Procedure: FDG-PET scan — imaging scan
  Groups: 2

SUMMARY:
A study to determine the accuracy of FLT-PET in quantifying tumor cell proliferation at the initial staging of patients with Non-Hodgkin's Lymphoma in comparison wit the "gold standard" FDG-PET.

DETAILED DESCRIPTION:
The first primary objective reflects a necessary and preliminary requirement: to reproduce published results and validate the use of FLT-PET. In this study, 35 patients will be selected to undergoing imaging with both FLT and FDG PET.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Women must not be pregnant or breast feeding
* Histologic diagnosis of non-Hodgkin's lymphoma (any stage)
* Must undergo treatment with chemotherapy and/or radiotherapy

Exclusion Criteria:

* May not have received previous therapy with radiopharmaceuticals
* May not have received prior therapy with cytotoxic chemotherapy and/or monoclonal antibodies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects diagnosed with lymphoma and are about to start treatment with chemotherapy
Sampling Method: Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2008-10

PRIMARY OUTCOMES:
Staging and ReStaging scans | after hematopoetic recovery

CONTACTS AND LOCATIONS:
Locations (1):
- University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma, United States